CLINICAL TRIAL: NCT02508506
Title: A Phase 1 Study of the Pharmacokinetics, Safety, and Tolerability of ALKS5461 in Subjects With Renal Impairment
Brief Title: Pharmacokinetics and Safety of ALKS 5461 in Subjects With Renal Impairment and Normal Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALKS5461-A108
Record Dates: First submitted 2015-07-23; First posted 2015-07-27 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Renal Impairment
Keywords: ALKS 5461; Alkermes; Samidorphan; Renal Impairment; Pharmacokinetics; Buprenorphine
MeSH Terms: conditions — Renal Insufficiency | interventions — ALKS 5461

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ALKS 5461 (Experimental): Sublingual tablet
  Interventions: Drug: ALKS 5461

INTERVENTIONS:
Drug: ALKS 5461 — Single dose, given orally

SUMMARY:
This study will evaluate the effect of various degrees of renal function on the pharmacokinetics and safety of ALKS 5461.

ELIGIBILITY:
Inclusion Criteria:

For all subjects:

* Has a body mass index (BMI) of 18.0-40.0 kg/m^2 and a total body weight >50kg
* Agrees to use an approved method of contraception for the duration of the study
* Additional criteria may apply

For subjects with renal impairment:

* Has severe or end stage renal disease, and does not require dialysis
* Has stable renal function for at least 60 days preceding screening
* Additional criteria may apply

Exclusion Criteria:

For all subjects:

* Has any past history or current finding of a clinically significant observed abnormality, psychiatric or medical condition other than renal impairment
* Has a history of gastrointestinal surgery affecting drug absorption or biliary elimination, excluding appendectomy or cholecystectomy
* Is pregnant, planning to become pregnant, or lactating
* Has a history of clinically significant allergy or a hypersensitivity to opioids
* Additional criteria my apply

For subjects with renal impairment:

* Has evidence of compromised respiratory function, seizure disorder, or myasthenia gravis
* Has received a kidney transplant
* Additional criteria may apply

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve from time 0 to infinity (AUC0-inf) following a single dose of ALKS 5461 | up to 168 hours postdose
Area under the plasma concentration versus time curve from time 0 to time of last measurable concentration (AUC0-last) following a single dose of ALKS 5461 | up to 168 hours postdose
Maximum observed plasma concentration (CMAX) following a single dose of ALKS 5461 | up to 168 hours postdose

SECONDARY OUTCOMES:
Time to reach maximum plasma concentration (TMAX) | up to 168 hours postdose
Terminal elimination half-life (T1/2) | up to 168 hours postdose
Apparent clearance (CL/F) | up to 168 hours postdose
Apparent volume of distribution (Vz/F) | up to 168 hours postdose
Safety: Incidence of adverse events (SAE) | Up to 12 days

CONTACTS AND LOCATIONS:
Overall Officials: Arielle Stanford, MD, Study Director — Alkermes, Inc.
Locations (3):
- United States (3):
  - Alkermes Investigational SIte, Denver, Colorado
  - Alkermes Investigational SIte, Orlando, Florida
  - Alkermes Investigational Site, Minneapolis, Minnesota